CLINICAL TRIAL: NCT03931499
Title: Biochemical Predictors of Delirium in Patients Undergoing Cardiac Surgery Under Cardiopulmonary Bypass
Brief Title: Biochemical Predictors of Delirium in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Novosibirsk State University (Other)
Responsible Party: Sponsor
Other Study IDs: DEL2019
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Patients undergoing surgery under cardiopulmonary bypass
  Interventions: Diagnostic Test: Metabolomic analysis

INTERVENTIONS:
Diagnostic Test: Metabolomic analysis — Blood will be collected in all patients blood before surgery and after surgery (postoperative day 1). Our study is based on a polar metabolomics profiling of plasma and/or serum using hybrid triple quadrupole mass spectrometer coupled with chromatographic system.

SUMMARY:
Delirium is a common neurologic complication after cardiac surgery occuring in 30-50% of patients. The occurence of this complication is associated with worse outcomes, including prolonged length of stay in the ICU and hospital, increased morbidity and mortality. Considering great clinical significance of this complication, the search for early predictors of postoperative delirium remains an urgent task. The purpose of this prospective observational study is to test the hypothesis that metabolomic changes before and after cardiac surgery could be served as early predictors of this complication.

ELIGIBILITY:
Inclusion Criteria:

* surgery under cardiopulmonary bypass
* Age > 60 years
* CABG surgery or valve surgery (repair/replacement)

Exclusion Criteria:

* urgent surgery
* surgery on aorta
* combined procedures (CABG+valves)
* significant stenosis of carotid arteries
* Parkinson's disease
* liver cirrhosis
* use of anticholinergic drugs, antidepressants, antiepileptic or chemotherapy drugs

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing cardiac surgery under cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | 5 days after surgery
  Postoperative delirium will be diagnosed with CAM-ICU (confusion assessment method - intensive care unit)

CONTACTS AND LOCATIONS:
Locations (1):
- E. Meshalkin National Medical Research Center, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No